CLINICAL TRIAL: NCT05153902
Title: Impact of Regional Anesthesia on Blood Pressure in Humeral Fracture Surgery : Comparative Study Using Propensity-score
Brief Title: Impact of Regional Anesthesia on Blood Pressure in Humeral Fracture Surgery
Acronym: ALR_HUMERUS
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0647
Record Dates: First submitted 2021-10-19; First posted 2021-12-10 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Proximal Humeral Fracture
Keywords: Surgery; General Anesthesia; Regional anesthesia; Hypotension
MeSH Terms: conditions — Shoulder Fractures; Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to compare the hemodynamic impact of two anaesthetic strategies : Regional anesthesia versus General anesthesia in proximal humeral fracture surgery.

DETAILED DESCRIPTION:
Proximal humeral fracture surgery is frequently performed under General Anesthesia (GA).

GA is frequently associated with a high risk of hypotension with significant consequences.

Regional anesthesia could be an interesting alternative to GA in order to limit hemodynamic consequences, especially in elderly patients. Furthermore, in the current state of Covid 19 crisis, regional anesthesia could provide solutions in exposing less medical staff on patient's airway.

The investigators hypothesize that the use of Regional anesthesia reduces the use of intraoperative vasopressor during surgery.

After ethical committee approval, a retrospective cohort of patients with proximal humeral fracture, in Montpellier's University Hospital, was analyzed from 2016 to 2020. An informational note was given to all patients participating to the study.

ELIGIBILITY:
Inclusion Criteria:

* ASA I - IV
* Proximal humeral fracture
* Operated between january 2016 and december 2020
* Emergency surgery

Exclusion Criteria:

* Surgical revision or surgery for pre-existing infection, tumour
* Intubated patient / unconscious patient
* Haemostasis disorder
* Haemostasis disorder
* Refusal of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgery for Proximal humeral fracture between january 2016 and december 2020
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants requiring vasopressors in peroperative | during surgery (between anaesthethic induction and end of surgical procedure)
  Number of Participants who used vasopressors in peroperative

SECONDARY OUTCOMES:
Total dose of vasoconstrictor | during surgery (between anaesthethic induction and end of surgical procedure)
  Total dose of vasoconstrictor
Total time spent on vasopressor | during surgery (between anaesthethic induction and end of surgical procedure)
  Total time spent on vasopressor
Intraoperative complications | during surgery (between anaesthethic induction and end of surgical procedure)
  Intraoperative complications other than hypotension
Postoperative complications | between surgery and 2 days post-operative
  nausea/vomiting; cardiovascular complications; complications related to regional anesthesia ; postoperative cognitive disorders
total dose of rescue analgesia | between discharge from operating room and 24h post-operative
  opioids
Total time spent in the operating room | between arrival in the operating room and discharge from the operating room
  Total time spent in the operating room
Length of stay in duty or ICU | between the day of surgery and up to 1 month
  Length of stay in duty or ICU

CONTACTS AND LOCATIONS:
Locations (1):
- Uh Montpellier, Montpellier, France